CLINICAL TRIAL: NCT00885651
Title: A Randomised, Double Blinded, Crossover Study of the Influence of Metoprolol on Exercise Induced Elevation of Catecholamines in Healthy Subjects.
Brief Title: Ability of Metoprolol to Alter the Exercise Induced Elevation of Catecholamines
Acronym: MEXICHO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Morten Petersen, Department of Clinical Pharmacology, Rigshospitalet, Denmark, Morten Petersen, Department of Clinical Pharmacology, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-5-23-9-3-8-15; EudraCTnr. 2008-001908-23
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Heart Failure
Keywords: SNP; catecholamines; metoprolole; healthy subjects; physiological stress
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Metoprolol for 10 days followed by placebo for 7 days.
  Interventions: Drug: Metoprolole (Selo-Zok ®); Drug: Placebo
- 2 (Placebo Comparator): Placebo for 7 days followed by Metoprolol for 10 days
  Interventions: Drug: Metoprolole (Selo-Zok ®); Drug: Placebo

INTERVENTIONS:
Drug: Metoprolole (Selo-Zok ®) — Tablets, 200 mg, once a day, 10 days
Drug: Placebo

SUMMARY:
Heart failure is a frequent disease in Denmark, and it is associated with very high mortality. Around 60,000 people in Denmark have heart failure, and there is about 11,000 hospitalizations every year due to this disease. From the time of diagnosis, patients survive an average of 4-5 years.

A critical illness mechanism in heart failure is that these patients have high blood levels of catecholamines; epinephrine and norepinephrine, which is stress hormones from the sympathetic nervous system. Standard treatment of heart failure is with the two medical preparations betablockers and ACE-inhibitors.

It is not known what effect betablocker-treatment have on blood concentration of epinephrine and norepinephrine.

It is the purpose of this study, to investigate the effect of Selo-Zok ® (metoprolol) on the blood concentration of epinephrine and norepinephrine. This is done by creating a stress condition for the body, in this case with the bicycle test, while doing blood samples to determine the concentration of catecholamines. This will be done by 1-week treatment of tablet Selo-Zok ® followed by 1-week treatment of placebo (a substance with no medical effect). Blood samples will be taken to determine small changes in inheritance material (DNA) in the form of point mutations also called single nucleotide polymorphisms, since these changes can affect how we respond to metoprolol treatment.

ELIGIBILITY:
Inclusion Criteria:

* Kaukaser
* Healthy men
* 18 years < age < 30 years
* Non-smoker
* 18 < BMI < 25
* No chronic diseases
* Motor-disability that disables completement of cardio-pulmonary exercise-test.

Exclusion Criteria:

* Alcohol abuse or any other abuse
* Intake of any narcotic drugs (example: cannabinoids, narcotics, stimulants of central nervous system, hypnotics, hallucinogenes)
* Any of following medication:

  * astmamedication
  * heartmedication
  * antihistamines
  * antipsycotics
  * NSAIDs
  * rifampicine
  * chinidine
  * glucocorticoids
* Abnormal ECG, particularly 2. or 3. degree AV-block, sinusbradycardia, sick sinusnode-syndrome, sign of heart failure or ischemia.
* Allergy or intolerance of metoprolole
* Lactoseallergy
* 110 mmHg < Systolic blood pressure < 140 mmHg
* 60 mmHg < Diastolic blood pressure < 90 mmHg
* Bloodsucker > 11,1 mmol/L, or fasting, venous bloodsucker >= 7,0 (measured if: 7,8 < BS < 11,1)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Changes in stress-triggered response of catecholamines. | 2 weeks and 3 days

SECONDARY OUTCOMES:
Change in stress-triggered blood pressure response. | 2 weeks and 3 days
Change in stress-triggered pulse response. | 2 weeks and 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Henrik HP Enghusen Poulsen, MD, Principal Investigator — Rigshospitalet, Universityhospital of Copenhagen

REFERENCES:
- [Derived] Petersen M, Andersen JT, Jimenez-Solem E, Broedbaek K, Hjelvang BR, Henriksen T, Frandsen E, Forman JL, Torp-Pedersen C, Kober L, Poulsen HE. Effect of the Arg389Gly beta(1)-adrenoceptor polymorphism on plasma renin activity and heart rate, and the genotype-dependent response to metoprolol treatment. Clin Exp Pharmacol Physiol. 2012 Sep;39(9):779-85. doi: 10.1111/j.1440-1681.2012.05736.x. PMID 22703382